CLINICAL TRIAL: NCT00198276
Title: An Open-Label Study Using the MedPulser Electroporation System to Treat Cutaneous and Subcutaneous Foci of Cancer
Brief Title: Study Using the MedPulser Electroporation System With Bleomycin to Treat Cutaneous and Subcutaneous Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU-CCBE-2003
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Cancer
Keywords: cancer; cutaneous; subcutaneous; MedPulser; bleomycin; electroporation; Cutaneous or subcutaneous cancer
MeSH Terms: conditions — Neoplasms | interventions — Bleomycin

STUDY DESIGN:
Intervention Model Description: MedPulser Electroporation with Belomycin
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bleomycin (Experimental): Bleomycin 4.0 U/mL at dose of 1 U/cm^3 of treatment area; Medpulser EP
  Interventions: Combination Product: MedPulser Electroporation with bleomycin

INTERVENTIONS:
Combination Product: MedPulser Electroporation with bleomycin — The MedPulser device will be used in combination with Bleomycin Sulfate injection around the tumor area in a concentration of 1 U/ml per cm3 of tumor treatment area.

SUMMARY:
The purpose of the study is to study the safety and efficacy of MedPulser Electroporation with bleomycin treatment of cutaneous and subcutaneous foci of cancer.

DETAILED DESCRIPTION:
Electroporation therapy (EPT) is a tumor-specific ablative treatment modality with the potential to manage local tumors without the potentially undesirable side effects of systemic chemotherapy agents or radiotherapy. Surgical resection of cutaneous lesions may lead to significant organ dysfunction and/or permanent disfigurement requiring reconstructive surgery (i.e. nose, eye area, ears, medial canthus, nasolabial fold, lip, scalp, etc.). In contrast, electroporation therapy may offer equivalent disease control to conventional surgery with a lessened need for reconstructive surgery.

The ability to ablate local cutaneous lesions with the MedPulser® System when used in conjunction with intralesional Bleomycin is an important new treatment for the local management of recurrent Basal Cell Carcinoma (BCC), recurrent Squamous Cell Carcinoma (SCC), Melanoma, Adenocarcinoma (i.e. local recurrence of breast cancer), Merkel Cell Carcinoma and Cutaneous Lymphoma and other solid tumors with symptomatic subcutaneous recurrences and provides an alternative treatment option to subjects who:

1. have failed standard treatments; or who
2. are unwilling or unsuitable to undergo conventional surgical excision or radiation.

EPT with Bleomycin spares normal tissue and its use in local disease management may preserve organ function and/or appearance relative to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of recurrent SCC, recurrent BCC, melanoma, adenocarcinoma (i.e., local recurrence of breast cancer), merkel cell carcinoma, cutaneous lymphoma, other subcutaneous solid tumors, or primary cutaneous tumors must be confirmed by histological examination of a tissue (e.g., biopsy) sample obtained within 1 month prior to a patient signing the informed consent form for the study.
2. Total volume of disease treated will require a dose of bleomycin sulfate less than 80 units.
3. Tumors and margins must be completely accessible to intralesional bleomycin injections and the EPT applicator electrodes.
4. Age: 18 years or older.
5. Male or female.
6. Men and women of childbearing potential must be using physician prescribed contraceptive methods while undergoing protocol related therapy.
7. Baseline performance status: ECOG 0-2

   * Grade 0: Fully active, able to carry on all pre-disease performance without restriction.
   * Grade 1: Restricted in a physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
   * Grade 2: Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours.
8. Life expectancy of at least 6 months.
9. Sign a written Informed Consent prior to receiving any study procedures or treatments.

Exclusion Criteria:

1. Subjects with tumors suspected of involving a 50% or greater encasement of a blood vessel as measured by magnetic resonance imaging (MRI) or computed tomography (CT) scan.
2. Subjects with tumors having bone invasion.
3. Subjects with hypersensitivity to bleomycin.
4. Subjects who have received or will exceed a total lifetime dose of bleomycin greater than 400 units.
5. Subjects with a significant history of emphysema or pulmonary fibrosis.
6. Subjects with indwelling cardiac pacemakers who cannot tolerate a period with pacemaker turned off.
7. Subjects with a history of uncontrolled cardiac arrhythmia.
8. Women who are pregnant, or are nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2004-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Local tumor control | 6 Months

SECONDARY OUTCOMES:
Pharmacoeconomic factors (e.g. hospital costs, extent of medical interventions, medication use) | 24 Months
MedPulser instrument and applicator performance | 6 Months
Adverse events | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Goldfarb, MD, Study Chair — Inovio Pharmaceuticals
Locations (1):
- Inovio Biomedical Corporation, San Diego, California, United States